CLINICAL TRIAL: NCT05295797
Title: The Positively Dance Pilot Program: Examining the Feasibility of a Peer Research Associate-Led Dance Program for Women Living With HIV
Brief Title: The Positively Dance Pilot Program for Women Living With HIV
Acronym: Dance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Simon Fraser University (Other)
Responsible Party: Principal Investigator, Eli Puterman, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H20-03483
Record Dates: First submitted 2022-03-02; First posted 2022-03-25 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; dance; peer-led
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Thirty WLWH will be enrolled and randomized to the (1) group-based 12-week dance program (N=15) or (2) waitlist control (N=15) (participants in the waitlist control will be assigned to a waiting list and will be invited to participate in dance classes after the intervention arm 12-week dance program has ended).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance Program (Experimental): Participants will take 2 in person dance classes led by peer dance instructors per week for 12 weeks
  Interventions: Behavioral: Dance Program
- Control (No Intervention): Participants in the waitlist control will be assigned to a waiting list and will be invited to participate in dance classes after the intervention arm 12-week dance program has ended

INTERVENTIONS:
Behavioral: Dance Program — Participants will take 2 in person dance classes led by peer dance instructors per week for 12 weeks
  Arms: Dance Program

SUMMARY:
The Positively Dance study involves the assessment of the accessibility and feasibility of a 12-week randomized aerobic dance pilot program that will provide women living with HIV with the opportunity to take part in dance classes with women living with HIV as the dance instructors.

DETAILED DESCRIPTION:
Women living with HIV (WLWH) are at greater risk of advanced cellular aging, comorbidities, and early mortality than men living with HIV or women in the general population. WLWH face significant social and economic disadvantages which serve as barriers to accessing HIV therapy or other programming that could support their health and wellbeing. It is thus critical to identify amenable healthy aging factors to ameliorate the burden of HIV for WLWH.

Aerobic training has consistently been shown to reduce disease risk and early mortality in the general population and in people living with HIV. Immune system function partly underlies many of the cardiovascular, lung, muscular, and neural benefits of aerobic exercise. While sporadic immune activation is typical during innate and adaptive immune responses, the development and pathogenesis of non-communicable diseases are now understood to result from chronic, low-grade, systemic inflammation in the body, known as inflamm-aging as seen among people living with HIV even when their viremia is controlled by therapy. Systemic inflammation results from multiple sources, including, but not limited to, accumulation of fat and immunosenescent cells, the latter of which no longer divide but secrete damaging inflammatory cytokines. Immunosenescent cells are marked by several biomarkers, though most attention has been directed towards average telomere lengths of immune cells. Telomeres are genepoor regions located at the ends of chromosomes and are formed by hexameric 5'(TTAGGG) n3' repeats and shortened telomeres portend earlier replicative senescence - when cells no longer replicate but live on in a pro-inflammatory state - or programmed cellular death. 24 weeks of physical activity is associated with apparent reversal of the aging process of immune cells with increases in average leukocyte (i.e. immune cells) telomere lengths (LTL).

While aerobic exercise benefits people living with HIV, a recent review emphasizes that WLWH and adults from minority groups are less likely to engage in or are more likely to withdraw from standard exercise programs. Consultations with The Canadian HIV Sexual and Reproductive Health Cohort Study (CHIWOS) Advisory Board of WLWH identified and prioritized the need for interventional research to mitigate the effects of accelerated aging and decrease the risk of disease, and identified dance as a particularly exciting program to study, if made free and easily accessible.

This study will be a 12-week randomized dance pilot program. The dance classes will be led by trained peer dance instructors who are also WLHIV.

Prior to consent, participants will be screened for inclusion/exclusion criteria. Next, participants will be invited to an in-person, paid orientation session to review study objectives and discuss the pros/cons to participating in the pilot program and randomization to either a waitlist control or active study arm. After consent, participants will then be asked to complete blood draws and a pre-intervention survey.

Each dance instructor (PRA) will lead 1-2 classes (50-min/class) per week (depending on availability) for 12 weeks, with an expectation that women in the pilot's active arm have access to 2 classes per week during the first 12 weeks of active data collection. Classes will be offered in person at a local dance studio. Attendance will be taken at each dance class by throughout the 12 weeks. Participants will also have the opportunity to socialize during breaks after dance classes for as long as they wish for up to half an hour.

Following the 12 weeks of active data collection for the pilot program, all participating women will be asked to return to complete blood draws and a repeat survey to collect post-intervention data on physical activity levels, mental and physical health, and social integration. We will also conduct semi-structured interviews with all women in the active arm to learn more about their experiences in and impressions of the program.

Our 12-week program will be followed by 12 more weeks of dance classes where waitlist women are invited to join the classes. Attendance of all women will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as women living with HIV
* Are over the age of 18
* Are able to speak and read English
* Are able and willing to commit to participating in dance classes 2 times a week per week for 12 weeks
* Be able to attend in person dance classes
* Meet minimal risk clearance to engage in exercise (screened with the Physical Activity Readiness Questionnaire PARQ+)

Exclusion Criteria:

* Do not self-identify as a woman living with HIV
* Are under the age of 18
* Cannot speak and read English
* Cannot attend in person dance classes
* Do not meet minimal risk clearance to engage in exercise (screened with the Physical Activity Readiness Questionnaire PARQ+)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman-identified
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of women who accept the invitation to participate in the research study | Throughout the recruitment phase, up to 1.5 months
  This information will be used to understand feasibility
Number of women who initially participate in the intervention | Week 1-12
  This information will be used to understand feasibility
Proportion of women who participate in the dance classes, even after the active data collection phase is completed | Week 13-24
  To determine the extent to which women continue attending the dance classes for an additional 12 weeks, if the classes are offered for free. This information will be used to understand feasibility.
Acceptability and feasibility of the selected procedures (e.g. blood draws, questionnaires) by determining numbers who attend these sessions and complete the questionnaires | Baseline (Week 0) and at the end of the program (Week 13)
  This information will be used to understand feasibility and acceptability
Adverse events that may occur during the trial | Week 1-24
  This information will be used to understand feasibility
Continued participation of the peer dance instructors | Week 1-24
  This information will be used to understand feasibility
Individual semi-structured interviews asking participants their perceptions of and experiences with the program | Once after Week 12, up to 4 weeks after
  To determine the accessibility and feasibility of the intervention, we will conduct individual semi-structured qualitative interviews with the participants who took part in the intervention arm of the study as well as with the peer dance instructors. The women will be asked about their perceptions of and experiences with the program, including why they joined the program, what they liked and disliked about the program, what the program meant to them, how effective they thought the program had been, what barriers to participation they faced throughout the intervention, and their suggestions for future program delivery. Interviews will occur via Zoom or in-person depending on the participant's preferences and will be audio-recorded (only the audio portion of the interviews will be recorded).

SECONDARY OUTCOMES:
Changes in whole blood telomere length | Baseline (Week 0) and at the end of the program (Week 13)
  Whole blood telomere length, using the standard approach of measuring relative telomere lengths with quantitative polymerase chain reaction.
Changes in depressive symptoms measured with the Patient Health Questionnaire-9 | Baseline (Week 0) and at the end of the program (Week 13)
  The Patient Health Questionnaire-9 (PHQ) is the self-administered depression module of the full Patient Health Questionnaire. It scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Changes in general physical and mental health measured with the 36-Item Short Form Survey | Baseline (Week 0) and at the end of the program (Week 13)
  The 36-Item Short Form Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures relying on self-reporting. Likert scales and yes/no options are used to assess function and well-being on this 36-item questionnaire.
Changes in social support measured with the MOS Social Support Scale | Baseline (Week 0) and at the end of the program (Week 13)
  The MOS Social Support Survey measures four dimensions of functional social support. It is a 19-item multidimensional, self-administered instrument. Questions are answered on a five-point scale ranging from "none of the time" to "all of the time," with higher values indicating more support.
Changes in social connectedness measured with the Social Connectedness Scale | Baseline (Week 0) and at the end of the program (Week 13)
  This scale assesses the degree to which individuals feel connected to others in their social environment. Items are scored from 1 (strongly disagree) to 6 (strongly agree). Items are summed and a higher score indicates more connectedness to others.
Changes in social cohesion measured with the Social Assurance Scale | Baseline (Week 0) and at the end of the program (Week 13)
  The Social Assurance Scale is a 6 point Likert scale. Items are added up for a total score, and a higher score indicates more connectedness to others.
Changes in HbA1c | Baseline (Week 0) and at the end of the program (Week 13)
  Information will be used to determine means and standard deviations for these traditional health markers
Changes in C-Reactive Protein | Baseline (Week 0) and at the end of the program (Week 13)
  Information will be used to determine means and standard deviations for these traditional health markers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Burchell AN, Raboud J, Donelle J, Loutfy MR, Rourke SB, Rogers T, Rosenes R, Liddy C, Kendall CE. Cause-specific mortality among HIV-infected people in Ontario, 1995-2014: a population-based retrospective cohort study. CMAJ Open. 2019 Jan 8;7(1):E1-E7. doi: 10.9778/cmajo.20180159. Print 2019 Jan-Mar. PMID 30622108
- [Background] Hogg RS, Eyawo O, Collins AB, Zhang W, Jabbari S, Hull MW, Lima VD, Ahmed T, Kendall CE, Althoff KN, Justice AC, Barrios R, Shoveller J, Montaner JSG; Comparative Outcomes And Service Utilization Trends (COAST) study. Health-adjusted life expectancy in HIV-positive and HIV-negative men and women in British Columbia, Canada: a population-based observational cohort study. Lancet HIV. 2017 Jun;4(6):e270-e276. doi: 10.1016/S2352-3018(17)30029-2. Epub 2017 Mar 3. PMID 28262574
- [Background] Scully EP. Sex Differences in HIV Infection. Curr HIV/AIDS Rep. 2018 Apr;15(2):136-146. doi: 10.1007/s11904-018-0383-2. PMID 29504062
- [Background] Kendall CE, Wong J, Taljaard M, Glazier RH, Hogg W, Younger J, Manuel DG. A cross-sectional, population-based study measuring comorbidity among people living with HIV in Ontario. BMC Public Health. 2014 Feb 13;14:161. doi: 10.1186/1471-2458-14-161. PMID 24524286
- [Background] Patterson S, Cescon A, Samji H, Chan K, Zhang W, Raboud J, Burchell AN, Cooper C, Klein MB, Rourke SB, Loutfy MR, Machouf N, Montaner JS, Tsoukas C, Hogg RS; CANOC collaboration. Life expectancy of HIV-positive individuals on combination antiretroviral therapy in Canada. BMC Infect Dis. 2015 Jul 17;15:274. doi: 10.1186/s12879-015-0969-x. PMID 26183704
- [Background] Heissel A, Zech P, Rapp MA, Schuch FB, Lawrence JB, Kangas M, Heinzel S. Effects of exercise on depression and anxiety in persons living with HIV: A meta-analysis. J Psychosom Res. 2019 Nov;126:109823. doi: 10.1016/j.jpsychores.2019.109823. Epub 2019 Sep 2. PMID 31518734
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] O'Brien KK, Tynan AM, Nixon SA, Glazier RH. Effectiveness of aerobic exercise for adults living with HIV: systematic review and meta-analysis using the Cochrane Collaboration protocol. BMC Infect Dis. 2016 Apr 26;16:182. doi: 10.1186/s12879-016-1478-2. PMID 27112335
- [Background] Franceschi C, Garagnani P, Parini P, Giuliani C, Santoro A. Inflammaging: a new immune-metabolic viewpoint for age-related diseases. Nat Rev Endocrinol. 2018 Oct;14(10):576-590. doi: 10.1038/s41574-018-0059-4. PMID 30046148
- [Background] De Francesco D, Wit FW, Burkle A, Oehlke S, Kootstra NA, Winston A, Franceschi C, Garagnani P, Pirazzini C, Libert C, Grune T, Weber D, Jansen EHJM, Sabin CA, Reiss P; the Co-morBidity in Relation to AIDS (COBRA) Collaboration. Do people living with HIV experience greater age advancement than their HIV-negative counterparts? AIDS. 2019 Feb 1;33(2):259-268. doi: 10.1097/QAD.0000000000002063. PMID 30325781
- [Background] Keating SM, Golub ET, Nowicki M, Young M, Anastos K, Crystal H, Cohen MH, Zhang J, Greenblatt RM, Desai S, Wu S, Landay AL, Gange SJ, Norris PJ; Women's Interagency HIV Study. The effect of HIV infection and HAART on inflammatory biomarkers in a population-based cohort of women. AIDS. 2011 Sep 24;25(15):1823-32. doi: 10.1097/QAD.0b013e3283489d1f. PMID 21572306
- [Background] Blackburn EH, Gall JG. A tandemly repeated sequence at the termini of the extrachromosomal ribosomal RNA genes in Tetrahymena. J Mol Biol. 1978 Mar 25;120(1):33-53. doi: 10.1016/0022-2836(78)90294-2. No abstract available. PMID 642006
- [Background] Moyzis RK, Buckingham JM, Cram LS, Dani M, Deaven LL, Jones MD, Meyne J, Ratliff RL, Wu JR. A highly conserved repetitive DNA sequence, (TTAGGG)n, present at the telomeres of human chromosomes. Proc Natl Acad Sci U S A. 1988 Sep;85(18):6622-6. doi: 10.1073/pnas.85.18.6622. PMID 3413114
- [Background] Campisi J, d'Adda di Fagagna F. Cellular senescence: when bad things happen to good cells. Nat Rev Mol Cell Biol. 2007 Sep;8(9):729-40. doi: 10.1038/nrm2233. PMID 17667954